CLINICAL TRIAL: NCT04201470
Title: Serum Neurofilaments Light Chain and GFAP (Glial Fibrillary Acidic Protein) in Atypical Idiopathic Inflammatory Demyelinating Disorders
Brief Title: Serum Neurofilaments and GFAP in Atypical Multiple Sclerosis
Acronym: AMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL17_0381
Record Dates: First submitted 2019-12-10; First posted 2019-12-17 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Progressive Multiple Sclerosis; Controls; Multiple Sclerosis
Keywords: Atypical multiple sclerosis; Cavitary multiple sclerosis; Myelocortical multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MS patients (Experimental): Patients with atypical MS identified in our cohort
  Interventions: Other: Blood withdrawal; Other: MRI; Other: Neurologic / neuropsychologic tests - Patients
- Controls (Active Comparator)
  Interventions: Other: Blood withdrawal; Other: MRI; Other: Neurologic / neuropsychologic tests - Controls

INTERVENTIONS:
Other: Blood withdrawal — Measurement of serum neurofilaments light chain and GFAP
Other: MRI — Cervical and cerebral MRI without contrast injection
Other: Neurologic / neuropsychologic tests - Patients — EDSS (Expanded Disability Status Scale), NHPT (Nine Hole Peg Test), T25FW (Timed 25-Foot Walk Test), 6MWT (Six-Minute Walk Test), CSCT (Computerized version of the Symbol Digit Modalities Test)
  Arms: MS patients
Other: Neurologic / neuropsychologic tests - Controls — NHPT, T25FW, CSCT
  Arms: Controls

SUMMARY:
Idiopathic inflammatory disorders of the central nervous system include various disorders of which multiple sclerosis is the most common. Besides multiple sclerosis, other distinct disorders including for example anti-AQP4 (aquaporine-4) and anti-MOG (Myelin oligodendrocyte glycoprotein) NMOSD (Neuromyelitis optica spectrum disorder) have been well characterized and are now known to be distinct from MS.

some patient belonging to MS spectrum have recently being characterized but unusual MRI findings have mimicking inherited leukoencephalopathies and leukodystrophies.

Whether these patients with atypical phenotype represent a separate disease distinct from MS or belong to MS spectrum is not clear.

The objectives are to evaluate a series of 15 patients with atypical forms of MS using non-conventional MRI techniques and biological biomarkers (serum neurofilaments light chain) and to compare them with classical MS patients (15 relapsing remitting patients and 15 progressive patients) and 15 controls. the hypothesize is that these patients with atypical MS have a more severe neurodegenerative process.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have given his informed consent and signed the consent form (if patient is protected by the law due to the study pathology, the consent will be signed his tutor or guardian ; if patient is unable to read or sign the consent form due to the study pathology, the consent will be signed by his family/trusted person)
* The subject is at least 18 years old (≥).
* Affiliate or beneficiary of a social security scheme

Inclusion criteria specific to Patients:

* Patients with atypical form of MS
* OR patients with RRMS (Relapsing-Remitting Multiple Sclerosis)
* OR patients with PPMS (Primary Progressive Multiple Sclerosis)

(Patients will be matched on EDSS score (+/-1) and age (+/-5) ; Controls will be matched with patients on age)

Exclusion Criteria:

* Pregnant or lactating women.
* Vulnerable people.
* Simultaneous participation in any other research protocol.
* Contraindication to the realization of an MRI (ferromagnetic ocular or cerebral foreign bodies close to nerve structures, pace-maker, cochlear implants)
* Claustrophobic subject
* Subject presenting a neurodegenerative disease (Parkinson, Alzheimer ...)
* Subject presenting psychiatric disorders like psychosis, excluding anxio-depressive episode
* Subject presenting a systemic pathology with neurological manifestation
* Subject presenting anterior or evolutionary neurological pathology other than the 3 entities defined in the inclusion criteria
* Subject presenting or having had a history of severe group 2 or 3 head trauma according to the Masters classification
* Patient receiving high dose corticosteroid therapy in the 3 months prior to inclusion in the study

Exclusion criteria specific to Patients:

* Patient who is taking, or who has taken in the last year, one of the following treatments: Fingolimod, or any Monoclonal Antibody (Natalizumab, Rituximab, Ocrelizumab, Alemtuzumab ...)
* Patient having had an outbreak of the disease in the 3 months prior to inclusion in the study

Exclusion criteria specific to Controls:

* Subjects who are protected or unable to give their consent
* Subject with anterior or progressive neurological pathology
* Patient being treated or having taken any Monoclonal Antibody
* In the period of exclusion relating to another protocol or for which the annual amount of the maximum indemnities of 4500 € has been reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Serum neurofilaments light chain | Between baseline (day 0) and day 60
  Evaluation of serum neurofilaments light chain levels in patients with atypical MS and comparison with controls and patients with classical MS

SECONDARY OUTCOMES:
Serum GFAP | Between baseline (day 0) and day 60
  Evaluation of serum GFAP levels in patients with atypical MS and comparison with controls and patients with classical MS

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No